CLINICAL TRIAL: NCT03125928
Title: Single Arm, Phase IIA Clinical Trial Assessing The Safety And Efficacy of Atezolizumab in Combination With Paclitaxel, Trastuzumab, and Pertuzumab in Patients With Metastatic HER-2 Positive Breast Cancer
Brief Title: Clinical Trial of Atezolizumab With Paclitaxel, Trastuzumab, and Pertuzumab in Patients With Metastatic HER-2 Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-093; 17-1010 (Other: Fox Chase Cancer Center IRB)
Record Dates: First submitted 2017-03-22; First posted 2017-04-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HER2-positive Breast Cancer
Keywords: Atezolizumab; PD-L1
MeSH Terms: interventions — atezolizumab; Paclitaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Arm (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Atezolizumab — Monoclonal antibody
Drug: Paclitaxel — Chemotherapy
Drug: Trastuzumab — Monoclonal antibody
Drug: Pertuzumab — Monoclonal antibody

SUMMARY:
This is a single arm, Phase IIA clinical trial assessing the safety and efficacy of atezolizumab in combination with paclitaxel, trastuzumab, and pertuzumab in 50 patients with locally advanced, unresectable, or metastatic HER2-overexpressing breast cancer. Due to concerns that corticosteroids may have a negative effect on tumor immunity expected with addition of atezolizumab to the standard of care regimen, patients will receive premedication with dexamethasone only for weeks 1 and 2 of the weekly paclitaxel, and then corticosteroid premedication will be discontinued subsequently.

Patients must have pathologically confirmed HER2-overexpressing breast cancer that is locally recurrent, unresectable, or metastatic, with measurable disease as defined by RECIST v1.1. Tumor measurements and bone scans will be performed every 9 weeks while patients are on study.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with pathologically confirmed HER2-overexpressing breast cancer, that is locally recurrent, unresectable or metastatic (negative or positive for ER/PR, and positive for HER2).
* HER2 status confirmed positive by means of immunohistochemistry (IHC) or in situ hybridization (ISH) according to ASCO/CAP 2013 guidelines. It is considered positive if scored as 3+ by an IHC method defined as uniform membrane staining for HER2 in 10% or more of tumor cells or demonstrate HER2 gene amplification by an ISH method (single probe, average HER2 copy number ≥ 6.0 signals/cell; dual probe HER2/CEP17 ratio ≥2.0 with an average HER2 copy number ≥4.0 signals/cell; dual probe HER2/chromosome enumeration probe (CEP)17 ratio ≥2.0 with an average HER2 copy number <4.0 signals/cell; HER2/CEP17 ratio <2.0 with an average HER2 copy number ≥ 6.0 signals/cell).
* Have measurable clinical disease: Measurable disease, defined as at least 1 measurable lesion on a CT scan as defined by RECIST (version v1.1).
* Age > 18 years.
* ECOG performance status 0,1or 2.
* Adequate organ function (defined by the following parameters): Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. Hemoglobin ≥ 10 g/dL.Platelets ≥ 100 x 109/L. Serum bilirubin ≤ 1.5 x upper normal limit (UNL), except patients with Gilbert's syndrome. Serum alanine aminotransferase (ALT) ≤ 2 x UNL or ≤ 5.0 x UNL in case of liver metastases. Serum aspartate aminotransferase (AST) ≤ 2 x UNL or ≤ 5.0 x UNL in case of liver metastases. Serum creatinine < 140 μmol/L (< 1.6 mg/dL) or 1.5x the upper limit of normal, whichever is less. Serum alkaline phosphatase (ALP) ≤ UNL or ≤ 2.5 x ULN in case of liver and bone metastases.
* Left ventricular ejection fraction of 50% or more at baseline (by echocardiography or multiple-gated acquisition scanning).
* Patients may have received one prior hormonal treatment for metastatic disease.
* Patients may have received adjuvant or neoadjuvant chemotherapy with or without trastuzumab and pertuzumab with an interval greater than than 12 months since completion of adjuvant/neoadjuvant treatment.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
* Female participants of childbearing age must be willing to use contraception methods, or abstain from sexual activity throughout the course of the study and for 7 months after the last dose of atezolizumab.
* Have provided tissue from a newly obtained biopsy obtained from a focus of metastatic disease, and be willing to consider repeat biopsy post-treatment after at least 4 cycles of treatment (an archival tissue sample may be substituted if new biopsy cannot be obtained and by discretion of Sponsor Investigator).

Exclusion Criteria:

* Patients participating in another trial of an investigational agent within 4 weeks of the 1st dose of the study.
* Patients with tumors that cannot be measured or clinically followed.
* Patients who had received therapy for metastatic breast cancer (other than that described above).
* Patients with active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 4 weeks prior to trial treatment.
* Patients with any baseline grade 2 neuropathy.
* Patients with known prior hypersensitivity reaction to any of the study drugs.
* Active autoimmune disease that is requiring systemic treatment within the past 3 months or documented history of clinically active autoimmune disease that requires systemic corticosteroids or immunosuppressive therapy.
* Diagnosis of immunosuppression or receiving steroid therapy or other immunosuppressive therapy within 4 weeks of the study.
* Have evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Patients with human immunodeficiency virus (HIV1/2). An HIV test must be performed to confirm status prior to enrollment.
* Patients who are carriers of hepatitis virus B and C. Hepatitis B and C testing must be performed to confirm status prior to enrollment.
* Prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death 1 ligand (PDL-1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte -associated antigen-4 (CTLA-4) antibody.
* Pregnant, breastfeeding, or expecting to conceive within the projected time of the trial, starting with the pre-screening or screening visit and through 7 months after the last dose of trial treatment.
* Active infection requiring systemic therapy.
* Active substance abuse or psychiatric disorders.
* The use of a RANKL inhibitor (denosumab) must be discontinued during the study. Bisphosphonate therapy is permitted.
* The following treatments must be discontinued: Herbal Medications. Immunomodulatory agents, including but not limited to interferons or IL-2. Immunosuppressive medications, including but not limited to cyclophosphamide, azathioprine, methotrexate, and thalidomide. Systemic corticosteroids. Anti-TNF-α agents.
* Any live, attenuated vaccine within 28 days prior to the first day of treatment or during study treatment, or unwillingness to avoid live, attenuated vaccines within 90 days following the last dose of atezolizumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Up to 5 years after stopping study treatment
  Treatment-related adverse events will be assessed by CTCAE v4.0
Antitumor activity of atezolizumab plus the standard regimen of paclitaxel, trastuzumab, and pertuzumab | An average of 18 weeks
  Antitumor activity will be measured by RECIST v1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after the last patient stops treatment
  OS is defined as the time from initiation of treatment until death from any cause or end of the study period, whichever occurs first.
Time to tumor progression (TTP) | Up to 5 years after the last patient stops treatment
  TTP is defined as the duration of time from the start of treatment to the first objectively documented instance of progressive disease.
Time to treatment failure (TTF) | Up to 5 years after the last patient stops treatment
  TTF is defined as the duration of time from start of treatment to discontinuation of study treatment for reasons defined in the protocol.
Progression free survival (PFS) | Up to 5 years after the last patient stops treatment
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Clinical benefit rate (CBR) | Up to 5 years after the last patient stops treatment
  CBR is defined as the rates of complete response (CR), partial response (PR) and stable disease (SD).
Duration of response (DOR) | Up to 5 years after the last patient stops treatment
  Per RECIST v1.1, DOR will be assessed by the duration of overall response, duration fo CR/PR, and duration of SD.
Correlation of biomarkers related to PD-L1 blockade with objective response rate (ORR), CBR, PFS, OS, and DOR. | Up to 5 years after the last patient stops treatment
  Efficacy will be assessed according to tumor PD-L1 expression level and tumor infiltrating lymphocytes PD-L1 expression levels.
Efficacy according to hormone receptor status (ER/PR) | Up to 5 years after the last patient stops treatment
  This will be a future subset analysis.
Feasibility of discontinuation of corticosteroids use after 2 weekly doses of paclitaxel | Up to 5 years after the last patient stops treatment
  This will be assessed by CTCAE v4.0.
Rate of occurrence of paclitaxel-related infusion hypersensitivity reaction after discontinuation of corticosteroids | An average of 18 weeks
  This will be assessed by CTCAE v4.0.
Cardiac safety | An average of 18 weeks
  Quarterly MUGA or ECHO results assessing occurrence of left ventricular dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States